CLINICAL TRIAL: NCT07230951
Title: Interaction Between White Potato Consumption and Meal Timing on Glycemic Response, Subjective Appetite, and Energy Intake in Adults.
Brief Title: Interaction Between White Potato Consumption and Meal Timing on Glycemic Response and Appetite in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, PhD, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: REB: 25-172 [A]
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy; Adult; Appetite; Glycemic Response; Mealtiming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Oven-baked Home Fries (Experimental): Test Treatment
  Interventions: Other: Oven-baked Home Fries
- Oven-baked White Russet Potato (Experimental): Test Treatment
  Interventions: Other: Oven-baked White Russet Potato
- Oven-baked Fries (Experimental): Test Treatment
  Interventions: Other: Oven-baked Fries
- Deep Fried, Quick Serve Fries (Experimental): Test Treatment
  Interventions: Other: Deep Fried, Quick Serve Fries
- Oven-baked Cauliflower Veggie Tots (Experimental): Test Treatment
  Interventions: Other: Oven-baked Cauliflower Veggie Tots
- No Side (Experimental): Test Treatment
  Interventions: Other: No Side

INTERVENTIONS:
Other: Oven-baked Home Fries — Oven-baked Home Fries (241 g; McCain Ltd.). Test treatments matched for calories (284 kcal)
  Arms: Oven-baked Home Fries
Other: Oven-baked White Russet Potato — Oven-baked White Russet Potato (299 g). Test treatments matched for calories (284 kcal)
  Arms: Oven-baked White Russet Potato
Other: Oven-baked Fries — Oven-baked Fries (201 g; McCain Ltd.). Test treatments matched for calories (284 kcal)
  Arms: Oven-baked Fries
Other: Deep Fried, Quick Serve Fries — Deep Fried, Quick Serve Fries (108 g; McCain Ltd.). Test treatments matched for calories (284 kcal)
  Arms: Deep Fried, Quick Serve Fries
Other: Oven-baked Cauliflower Veggie Tots — Oven-baked Cauliflower Veggie Tots (186 g; Green Giant). Test treatments matched for calories (284 kcal)
  Arms: Oven-baked Cauliflower Veggie Tots
Other: No Side — No side control (no caloric contribution).
  Arms: No Side

SUMMARY:
The purpose of this study is to evaluate the interaction between white potato consumption and meal timing on glycemic response, subjective appetite, and energy intake in adults. The investigators hypothesize that white potatoes will modulate glycemic response, enhance satiety, and mitigate subsequent meal consumption and overall food intake when compared with meals containing low glycemic carbohydrates. Furthermore, they anticipate that the timing of white potato consumption will yield differential effects, with breakfast consumption exerting a more pronounced impact on satiety and subsequent food intake reduction compared to dinner consumption.

DETAILED DESCRIPTION:
A randomized within-subject repeated measures experiment will be used to study the interaction between white potato consumption and meal timing on glycemic response, subjective appetite, and energy intake in adults. In Experiment 1, participants will consume, in a random order on separate mornings, one of six test meals consisting of an egg omelette and a test side of: (1) Oven-baked home fries, (2) Oven-baked white russet potatoes, (3) Deep-fried, quick serve fries, (4) Oven-baked fries, (5) Oven-baked cauliflower tots, or (6) no side. Acute glycemic response and subjective appetite will be measured at baseline and over 120-mins post treatment consumption. At 120-min, food intake will be evaluated via an ad libitum lunch. Rest of day food intake and glycemic response will be collected until the participant goes to bed. Blood glucose measurements will be collected using the Dexcom G7 continuous glucose monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years
* within the healthy body weight range [body mass index (BMI) between 18.5 - 24.9 kg/m2].

Exclusion Criteria:

* have a previous diagnosis of diabetes and gastrointestinal, liver or kidney disease;
* have had a major medical or surgical event within the past 6 months;
* have had any significant weight fluctuation in the past 6-months;
* are taking medication that may influence dependent measures;
* are or have been on a diet within the past 6 months;
* skip breakfast or are unable to consume test treatment food.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Glycemic Response (Acute Phase) | Change from baseline (measured at baseline (0-minute), 15-minute, 30-minute, 60-minute, 90-minute, and 120-minute post-treatment consumption).
  Blood glucose (mmol/L). Blood glucose concentrations will be measured using a Dexcom G7 CGM system.
Rest-of-day Blood Glucose | Continuous measurements for 24 hours post-treatment consumption.
  Blood glucose (mmol/L). Rest-of-day blood glucose concentrations will be determined using a Dexcom G7 CGM system.
Ad Libitum Food Intake | At 120 minutes post-treatment consumption
  Lunch pizza meal. Food intake will be determined by weighing the meal before and after serving. The net weight of the test meal will be converted to calories.

SECONDARY OUTCOMES:
Subjective Appetite | Change from baseline (measured at baseline (0-minute), 15-minute, 30-minute, 60-minute, 90-minute, and 120-minute post-treatment consumption).
  A visual analogue scale (VAS) with four questions will be administered to assess desire to eat, fullness, hunger, and prospective food consumption. Individual questions will be used to form a composite score. Each VAS will be administered via a digital software application (Express VAS, Toronto, Ontario, Canada) on a Dell tablet where participants will place an 'X" on the VAS line (100 unit scale).
Rest-of-day Food Intake | For the rest of the day following test session completion (1 day)
  Participants will be sent home with a rest-of-the-day food intake recall sheet to record their snacks, meals, and beverages. Rest of day food log.
Subjective Emotions | Change from baseline (measured at baseline (0-minute), 15-minute, 30-minute, 60-minute, 90-minute, and 120-minute post-treatment consumption).
  A visual analogue scale (VAS) with thirteen questions will be administered to assess subjective emotions and mood (aggression, anger, excitement, disappointment, happiness, upset, frustration, alertness, sadness, tension, exhaustion, calmness, and sleepiness). Individual questions will be used to form a composite emotion score. Each VAS will be administered via a digital software application (Express VAS, Toronto, Ontario, Canada) on a Dell tablet where participants will place an 'X" on the VAS line (100 unit scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Urban Innovation (CUI-109), School of Nutrition, Toronto Metropolitan University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No